CLINICAL TRIAL: NCT00656149
Title: Outcome Evaluation of Exercise and Electrical Therapy for Quadriplegic Hand Function
Brief Title: In-home Telerehabilitation for Quadriplegic Hand Function
Acronym: SCI-IHT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: International Spinal Research Trust (Other); Alberta Heritage Foundation for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SCI-IHT; ISRT-G700000249 PY107
Record Dates: First submitted 2008-04-01; First posted 2008-04-10 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Spinal Cord Injury; Quadriplegia; Tetraplegia
Keywords: telerehabilitation; functional electrical stimulation; spinal cord injury; hand function rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telerehabilitation of hand function (Active Comparator): Intervention: for one hour per day participants perform exercise therapy on a home-based tele-rehabilitation workstation, the Rehabilitation Joystick for Computerized Exercise (ReJoyce) with which participants play computer games associated with activities of daily life. A remote therapist coaches each one-hour session over the Internet, with the use of the ReJoyce tele-rehabilitation system. Hand grasp-release is assisted with functional electrical stimulation (FES) triggered voluntarily by the participant with the use of a wireless earpiece with a sensor that detects toothclicks.
  Interventions: Procedure: Telerehabilitation of hand function
- Conventional exercise therapy (Active Comparator): Intervention: for one hour per day participants perform conventional range-of-motion tasks with a wristlet weight (20 min), precision tasks with a computer mouse (20 min) and receive cyclical electrical stimulation of hand muscles (20 with the use of the ReJoyce tele-rehabilitation min). A remote therapist coaches each one-hour session A remote therapist coaches each one-hour session over the Internet, with the use of the ReJoyce tele-rehabilitation system.
  Interventions: Procedure: Conventional exercise therapy

INTERVENTIONS:
Procedure: Telerehabilitation of hand function — 6 weeks, 1 hr/day FES-assisted exercise therapy on a workstation, supervised over the Internet.
  Other Names: In-home telerehabilitation; Functional electrical stimulation (FES); Intensive exercise therapy; Massed practice
  Arms: Telerehabilitation of hand function
Procedure: Conventional exercise therapy — For one hour per day subjects perform range-of-motion tasks with a wristlet weight (20 min), precision tasks with a computer mouse (20 min) and receive cyclical electrical stimulation of hand muscles (20 min).
  Other Names: In-home telerehabilitation; Therapeutic electrical stimulation (TES); Intensive exercise therapy; Massed practice
  Arms: Conventional exercise therapy

SUMMARY:
1. To evaluate improvements in hand function in stable, cervical spinal cord injured (SCI) subjects treated with functional electrical stimulation (FES)-assisted exercise;
2. To compare the information obtained from existing qualitative and quantitative hand function tests with newly developed tests of sensorimotor performance.

Hypotheses:

1. the performance of tasks representative of activities of daily living (ADL) will improve with daily tele-supervised exercise of the affected hand.
2. The improvements will be greater in one exercise protocol than the other, the protocols being a) FES-assisted exercise on a workstation, b) cyclical FES, weight training and precision tasks.
3. Scores derived from quantitative data obtained from sensors on the workstation will correlate with the qualitative scores of the primary outcome measure, the ARAT hand function test.

DETAILED DESCRIPTION:
Chronic C5, 6 or 7 SCI subjects who have sustained a cervical SCI resulting in complete or incomplete quadriplegia. Time since injury at least one year at time of entry to study. Subjects may have a complete or an incomplete injury but must demonstrate loss of finger grasp and release as well as loss of thumb lateral (key) pinch bilaterally or unilaterally. Subjects must be stable neurologically and medically, cognitively intact, and willing and able to attend the requisite appointments for participation in the study.

Two treatments, each delivered 1 hour per day, five days a week over six weeks are given in a randomized order.

Treatment A

Subjects perform 1 hour per day of FES-assisted hand exercises on an instrumented exercise workstation in their homes, supervised remotely over the Internet. Four manipulanda in the workstation are used per exercise session. Each manipulandum is an object such as a spring-loaded doorknob, representing a task of daily life. As their motor skills improve over consecutive sessions, subjects are presented with manipulanda of increasing difficulty. A muscle stimulator garment is provided to each subject for FES-assisted exercise (Prochazka et al. 1997b). Hand opening and closing are wirelessly triggered from an earpiece that detects small voluntary tooth-clicks. The stimulator system is CSA-approved.

Treatment B Subjects perform the following tasks 1 hour per day in their homes, supervised remotely over the Internet.

1. 20 minutes of weight training: range of motion (ROM) movements while wearing a wristlet, the weight of which is selected so as to reduce the ROM at maximum effort by about 50%.
2. 20 minutes of accuracy training using a large computer mouse to play simple and enjoyable computer games that provide subjects with feedback on their performance.
3. 20 minutes of therapeutic electrical stimulation (TES). This consists of ON-OFF cyclical stimulation of hand muscles with the stimulator garment, e.g. while subjects watch TV.

The outcome measures are tested at 2-week intervals and require visits to the Center for Neuroscience at the University of Alberta. A maximum of CDN$2,000 is available to reimburse participants' travel and accommodation costs.

ELIGIBILITY:
Inclusion Criteria:

* Chronic C5, 6 or 7 SCI subjects who have sustained a cervical SCI resulting in complete or incomplete quadriplegia. Time since injury at least one year at time of entry to study. Subjects may have a complete or an incomplete injury but must demonstrate loss of finger grasp and release as well as loss of thumb lateral (key) pinch bilaterally or unilaterally. Subjects must be stable neurologically and medically, cognitively intact, and willing and able to attend the requisite appointments for participation in the study.

Exclusion Criteria:

* Subjects with unresolved medical issues such as easily triggered autonomic dysreflexia and/or hypotension.
* Subjects demonstrating severe spasticity affecting the upper extremities, fixed hand contractures with loss of suppleness and range of movement at the metacarpal-phalangeal joints, absence of voluntary ability to extend the wrist against gravity and/or insufficient muscle strength to abduct (lift) the arm against gravity.
* Subjects with unresolved substance abuse problems
* Subjects with a history of head injury, epilepsy in self or close relative and/or cognitive impairment
* Subjects with intracranial metal inclusions
* Subjects, who upon initial testing, demonstrate partial or complete denervation (loss of nerve supply) of the nerves to the the targeted muscle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test | every 2 weeks during therapy

SECONDARY OUTCOMES:
Transcranial magnetic stimulation | every 2 weeks during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Prochazka, Principal Investigator — University of Alberta
Locations (1):
- Centre for Neuroscience, University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Kowalczewski J, Chong SL, Galea M, Prochazka A. In-home tele-rehabilitation improves tetraplegic hand function. Neurorehabil Neural Repair. 2011 Jun;25(5):412-22. doi: 10.1177/1545968310394869. Epub 2011 Mar 3. PMID 21372246